CLINICAL TRIAL: NCT07084948
Title: Composition for Treating Acute Hepatitis, Chronic Hepatitis, Cirrhosis, and Hepatocellular Carcinoma for Hepatitis B Virus (SB Flavon)
Brief Title: Using Flavonoids to Kill Hepatitis B Virus
Acronym: Flavonoids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Trieu, Nguyen Thi, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SB Flavon
Expanded Access: NCT01198860 (Approved for marketing)
Record Dates: First submitted 2025-07-03; First posted 2025-07-25 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Hepatitis B Virus Infection
Keywords: Acid Ascorbic; L-Arginine hydrochloride; Urinariaflavone; 5,6-dihydroxy-7,8,4'-trimethoxy-flavone; Quercetin; Rutin; Kaempferol
MeSH Terms: conditions — Hepatitis B | interventions — Flavonoids; Tenofovir

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tenofovir 300mg + SB Flavon (Experimental): Experimental benefits in resistance to the Hepatitis B Virus were observed in all patients who had previously received certain components of the treatment for acute hepatitis, chronic hepatitis, cirrhosis, and hepatocellular carcinoma to Tenofovir + SB Flavon for various therapeutic purposes.
  Interventions: Drug: Flavonoid; Drug: Tenofovir
- Tenofovir 300mg (Experimental): Experimental benefits in resistance to the Hepatitis B Virus were observed in all patients who received the treatment with only Tenofovir for various therapeutic purposes.
  Interventions: Drug: Tenofovir

INTERVENTIONS:
Drug: Flavonoid — The daily maintenance, Tenofovir 150mg + SB Flavon 1345mg dose is to be taken 2 times a day, 1 tablet each time.
  The composition treats acute hepatitis, chronic hepatitis, cirrhosis, and hepatocellular carcinoma at an early stage. The product is Acid ascorbic, L-Arginine hydrochloride, Kaempferol, Urinariaflavone, 5,6-dihydroxy-7,8,4'-trimethoxy-flavone, Quercetin, Rutin.
  Use these ingredients to protect liver cell membranes, preventing the growth of HBV in the body.
  Other Names: Tenofovir + SB Flavon
  Arms: Tenofovir 300mg + SB Flavon
Drug: Tenofovir — The daily maintenance, Tenofovir 300mg dose is to be taken 1 time a day, 1 tablet each time.
  The composition treats acute hepatitis, chronic hepatitis, cirrhosis, and hepatocellular carcinoma.

SUMMARY:
The composition treats Acute Hepatitis, Chronic Hepatitis, Cirrhosis, and hepatocellular carcinoma (S.B.Flavonoids) at an early stage. The product is ascorbic acid, L-Arginine hydrochloride, Kaempferol, Urinariaflavone, 5,6-dihydroxy-7,8,4'-trimethoxy-flavone, Quercetin, and Rutin.

These components have participated in protecting liver cell membranes, focusing on reducing liver stress and supporting their structure, repairing and regenerating new liver parenchyma, preventing fibrosis cell generation, and preventing liver cancer cell growth at an early stage. The composition supplements precursors that help the body strengthen antibodies and reduce the risk of inflammation, and restore the physiological and biochemical functions of liver cells after chronic inflammation.

DETAILED DESCRIPTION:
The product is Acid ascorbic, L-Arginine hydrochloride, Kaempferol, Urinariaflavone, 5,6-dihydroxy-7,8,4'-trimethoxy-flavone, Quercetin, Rutin as the key compounds in the regeneration of to protect liver cell membranes, focus on reducing liver stress and supporting their prevent structure, fibrosis liver cell fibrosis, removing scar tissue, stimulate and release growth hormones, prevent progression to HCC, and prevent HCC recurrence.

The pharmaceutical ingredients involved in the composition are calculated to increase their effectiveness in preventing and curing acute hepatitis, chronic hepatitis, cirrhosis, and hepatocellular carcinoma.

Currently, many preparations have been and are being studied to fight against acute hepatitis, chronic hepatitis, cirrhosis, and liver cancer globally. The effectiveness of this preparation is a new finding that has been proven over 8 years of follow-up.

This ingredient is used as a supplement to stabilize the endothelium, regulate the amount of cortisol within normal limits, and help the body produce B lymphocytes with a good response.

Acid ascorbic, L-Arginine hydrochloride, Kaempferol, Urinariaflavone, 5,6-dihydroxy-7,8,4'-trimethoxy-flavone, Quercetin, Rutin. Flavonoids participate in cell protection against toxic proteins, which are produced during prolonged inflammation, blocking the action and removing denatured proteins that change the parenchyma of liver cells. The selected flavonoids repaired the fibrotic structure of liver parenchyma after chronic inflammation. Ascorbic acid and L-arginine help to facilitate biological functions in cell adhesion, synergize with flavonoids in cell membrane protection, structural repair, and liver cell regeneration.

ELIGIBILITY:
Inclusion Criteria:

* All patients with underlying medical conditions who have been taking medications for these conditions.
* Patients with AIDS, HIV, HBV, HCV, and patients with co-infections.
* The cancer patients are stable.
* Patients with congenital or acquired immunodeficiency.

Exclusion Criteria:

* Unstable cancer patients.
* Decompensated cirrhosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Quantification of HBV-DNA, SGPT, SGOT. The test uses sound waves to measure the stiffness of liver tissue on patient cirrhosis | 36 months
  HBV injure healthy liver cells, causing cell death and inflammation. Healthy liver tissue is replaced with scar tissue and the liver is damaged.

SECONDARY OUTCOMES:
The test uses sound waves to measure the stiffness of liver tissue on patient cirrhosis/Hcc (Arm 2) | 36 months
  Quantification of HBV-DNA, SGPT, SGOT. The test uses sound waves to measure the stiffness of liver tissue on patient cirrhosis carcinoma occurs most often in people with chronic liver diseases, cirrhosis, such as cirrhosis caused by hepatitis B.

CONTACTS AND LOCATIONS:
Locations (2):
- Saigon Biopharma LLC, Wilmington, Delaware, United States
- Saigon Biopharma Company Limited, Hồ Chí Minh, Ho Chi Minh City, Vietnam